CLINICAL TRIAL: NCT05165784
Title: Comparison of the Accuracy Between Technique V and Arterial Palpation Techniques in Determining the Location of the Femoral Veins
Brief Title: Comparison of Techniques in Determining Femoral Veins Location
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes123
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Vascular Access Complication
Keywords: arterial palpation technique; femoral access; femoral vein; V tecnique; vascular access

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- V technique (Active Comparator): Researcher will perform the V tecnique on the patient's inguinal area
  Interventions: Procedure: femoral vein identification
- palpation tecnique (Active Comparator): Researcher will perform the V tecnique on the patient's inguinal area
  Interventions: Procedure: femoral vein identification

INTERVENTIONS:
Procedure: femoral vein identification — Femoral vein identification using V technique
Procedure: femoral vein identification — Femoral vein identification using palpation technique

SUMMARY:
This study aimed to determine the accuracy of the V technique in predicting the location of the femoral vein compared to the technique of palpating the femoral artery with the use of USGss as a standard in determining the exact location of the femoral vein.

DETAILED DESCRIPTION:
One hundred and fifteen subjects were allocated into two large groups, V tecnique group and palpation tecnique group. Researchers will perform the V technique on the patient's inguinal area. This technique was performed using the researcher's contralateral hand. After the V technique is performed, the next researcher will perform the technique of palpating the femoral artery pulse at the exact location as the V technique. This technique is done by palpating the femoral artery pulsation using the examiner's index and middle fingers along the inguinal ligament; the location of the femoral vein is at 1 cm. medial to the femoral artery 2 cm inferior to the inguinal ligament. This location is marked "y" with a UV marker. researchers will compare the accuracy of both techniques in determining the exact location of femoral veins.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-65 years
* body mass index (BMI) of 18-25 kg/m2

Exclusion Criteria:

* could not lie supine
* had congenital or acquired abnormalities in the pelvic and inguinal region
* had a history of previous femoral vein puncture
* allergic to USG gel

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
prediction of femoral vein location | intra procedural
  Researcher will identify femoral vein location

CONTACTS AND LOCATIONS:
Overall Officials: Aida Rosita R Tantri, Doctor, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided